CLINICAL TRIAL: NCT02059564
Title: A Phase 1b, Exploratory, Randomized, Partially Single Blinded, Placebo and Open Label Controlled, Parallel Group Study to Assess the Effects of HM11260C and an Active Comparator on Gastric Emptying and Beta-Cell Response in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Phase 1b Study of LAPS-Exendin in Subjects of Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-EXC-102
Record Dates: First submitted 2014-02-05; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Exendin-4
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — Saline Solution; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): The weekly treatment of the 6 mg HM11260C or placebo will be maintained
  Interventions: Drug: HM11260C; Drug: Placebo
- Cohort B (Experimental): The monthly treatment with 4 mg HM11260C or placebo will be up titrated to 16 mg
  Interventions: Drug: HM11260C; Drug: Placebo
- Cohort C (Experimental): The daily treatment with 0.6 mg Victoza will be up titrated to 1.2 mg
  Interventions: Drug: Victoza

INTERVENTIONS:
Drug: HM11260C — doses of 6 mg, 16 mg
  Other Names: LAPS-Exendin-4
  Arms: Cohort A; Cohort B
Drug: Placebo — Normal saline solution
  Other Names: Normal saline solution
  Arms: Cohort A; Cohort B
Drug: Victoza — doses of 1.8 mg
  Other Names: Liraglutide
  Arms: Cohort C

SUMMARY:
A Phase 1b, Exploratory, Randomized, Partially Single Blinded, Placebo and Open Label Controlled, Parallel Group Study to Assess the Effects of HM11260C and an Active Comparator on Gastric Emptying and Beta-Cell Response in Subjects with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
Primary Objective

- effect of multiple different weekly and monthly doses of HM11260C and liraglutide (Victoza) as active control on gastric emptying

Secondary Objectives

* evaluate the pharmacodynamic (PD) effects of multiple weekly and monthly doses of HM11260C and liraglutide after a Mixed Meal Tolerance Test
* evaluate the islet β-cell function after a graded glucose infusion (GGI) of different doses of HM11260C and liraglutide
* evaluate safety and tolerability of different doses of HM11260C and liraglutide
* evaluate the pharmacokinetic (PK) effect of multiple weekly and monthly doses of HM11260C

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 to ≤ 70 years of age at the time of the Screening Visit
* History of type 2 diabetes
* Body mass index (BMI) ≥18 to ≤45 kg/m2 at the Screening Visit
* Use of approved methods of contraception
* Ability to provide written informed consent

Exclusion Criteria:

* Type 1 diabetes
* Significant acute diabetic proliferative retinopathy or severe neuropathy
* Systolic blood pressure >160 mm Hg and/or diastolic blood pressure >100 mm Hg at screening
* Pregnant or lactating women
* Participation in an investigational study within 30 days prior to randomization
* History of any major surgery within 6 months prior to Screening
* History of any serious adverse reaction or hypersensitivity to any of the product components.
* History of renal disease or significantly abnormal kidney function tests at Screening
* History of hepatic disease or significantly abnormal liver function tests
* History of any active infection within 30 days prior to Randomization
* Presence of clinically significant physical, laboratory, or ECG findings at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results
* Concurrent conditions that could interfere with safety and/or tolerability measurements per the investigator
* Donation or loss of >500 mL of blood or blood product within 56 days of Randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
PK profile of acetaminophen | 13 weeks
  Cmax, AUC at 13 weeks

SECONDARY OUTCOMES:
Glucose metabolism | 13 weeks
  Fasting plasma glucose (FPG), Postprandial glucose (PPG), Insulin, C-peptide, HbA1c at 13 weeks
Safety and tolerability | 18 weeks
  Incidence and severity of adverse events, findings on physical examination, clinical laboratory abnormalities at 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Clinical, Principal Investigator — California, United States
Locations (1):
- Hanmi, California City, California, United States

REFERENCES:
- [Derived] Hompesch M, Kang J, Han O, Trautmann ME, Sorli CH, Ogbaa I, Stewart J, Morrow L. Effects of efpeglenatide versus liraglutide on gastric emptying, glucose metabolism and beta-cell function in people with type 2 diabetes: an exploratory, randomized phase Ib study. BMJ Open Diabetes Res Care. 2021 Jun;9(1):e002208. doi: 10.1136/bmjdrc-2021-002208. PMID 34172436